CLINICAL TRIAL: NCT04043169
Title: Clearblue Pregnancy Test - Lay User Study
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-0971
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine sample Serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Clearblue pregnancy test — Urine pregnancy test

SUMMARY:
The Clearblue home pregnancy test (HPT) is an over-the-counter urine hCG (human chorionic gonadotropin) integrated digital test which is intended for the detection of pregnancy. This study will assess the performance of a HPT in the hands of lay-users by comparing their results when used according to the instructions for use (IFU) to (i) confirmed pregnancy status of the volunteers and (ii) to the results of trained study staff testing the same urine samples.

DETAILED DESCRIPTION:
The Clearblue product is an over-the-counter urine hCG (human chorionic gonadotropin) integrated digital test which is intended for the detection of pregnancy. The test is indicated for use from 6 days before the day of the missed period (5 days before the day of the expected period). The test is intended for home use.

This study aims to demonstrate that the Pregnancy Test has the required performance characteristics in lay-user testing, and when testing samples provided by lay-users. The study will recruit a cross-section of the target pregnancy test user population, that is, women aged between 18 and 45 representative of the intended user.

A minimum of 204 volunteers will be required to complete the study. The study site will aim to recruit an equal number of pregnant and not-pregnant volunteers (a minimum of 102 of each). Each volunteer will conduct the pregnancy test using both the 'in stream' and 'dip' method of sampling. Volunteer results will be evaluated against confirmed pregnancy status.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 to 45
* Willing to conduct a pregnancy test to determine or confirm their pregnancy status
* Willing to reveal their pregnancy status
* Willing to provide a blood sample
* Willing to give informed consent

Exclusion Criteria:

* Significant affiliation with SPD
* Has professional experience of using lateral flow-based devices
* Beyond the first trimester of pregnancy
* Taken a hormonal preparation containing hCG in the last month.
* Has a medical condition that means that it is not appropriate to give a blood.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female only
Study Population: Healthy pregnant, or not pregnant volunteers requiring or wishing to conduct a pregnancy test.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of Clearblue pregnancy test | 3 days
  Number of pregnancy test results in agreement with clinical pregnancy status

SECONDARY OUTCOMES:
Sample method agreement | 1 day
  number of volunteers who record the same pregnancy test result using the 'in stream' and 'dip' method of sampling
Coordinator agreement | 1 day
  number of volunteers who record the same pregnancy test result as a trained study coordinator
Device usability | 1 day
  number of volunteers who record the device as easy to use

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — SPD Development company Ltd.
Locations (1):
- WCCT, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided